CLINICAL TRIAL: NCT04729296
Title: Tumor Necrosis Factor Blocker (Anti-TNFα) to Delay or Prevent Progression to Stage 3 T1D
Brief Title: Anti-TNFα to Delay or Prevent Progression to Stage 3 T1D
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to COVID-19 related clinical limitations
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TN30 Anti-TNFα; 2U01DK106993-02 (NIH); 1UC4DK117009-01 (NIH)
Record Dates: First submitted 2021-01-20; First posted 2021-01-28 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — golimumab

STUDY DESIGN:
Intervention Model Description: Treatment assignment (active drug: placebo) will be assigned in a parallel, randomized, 1:1 model. Randomization will be conducted using block randomization with variable block sizes with stratification on TrialNet study site and age group (< 12 years old vs. 12 years old or older).
Who Masked: Participant, Investigator
Masking Description: Active drug and placebo will be identical in appearance and packaging
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Golimumab (Experimental): Golimumab for subcutaneous use
  Interventions: Drug: Golimumab
- Placebo (Placebo Comparator): Placebo syringes and vials matching active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Golimumab — For participants ≥45 kg, 50 mg of golimumab will be administered subcutaneously For participants <45 kg, the dose of golimumab is 30 mg/m2 to maximum of 50 mg
  Other Names: Simponi
  Arms: Golimumab
Drug: Placebo — Inactive Drug
  Arms: Placebo

SUMMARY:
This will be a study conducted as a placebo-controlled, double blind, 1:1 randomized controlled clinical trial testing a Tumor Necrosis Factor Blocker (Anti-TNFα) substance versus placebo in subjects with a 2-year 50% risk of progression to stage 3 T1D across multiple centers. The trial will investigate the ability of Anti-TNFα to prevent or delay progression to Stage 3 T1D in the targeted patient population.

ELIGIBILITY:
Inclusion Criteria:

Potential participants must meet all of the following inclusion criteria:

1. Age > 3 and < 46 years
2. Willing to provide Informed Consent or have a parent or legal guardian provide informed consent if the subject is <18 years of age
3. At least two or more diabetes-related biochemical autoantibodies insulin (mIAA), glutamic acid decarboxylase antibody (GADA), Islet cytoplasmic antibodies (ICA), islet antigen 2 (IA-2A), zinc transporter 8 (ZnT8A) present on the same sample. Of note, ICA and GADA positivity alone cannot be used to define eligibility in this trial).
4. Must have at least two of the high-risk markers defined below (within 7 weeks (52 days) of screening visit if performed as part of TN01 Pathway to Prevention (PTP) study at time of screening; defining a 50% two-year progression risk):

   a. Abnormal glucose tolerance: i. 2-hr glucose ≥ 140 and <200 mg/dL, fasting glucose ≥ 110 and <126, or 30-, 60-, or 90-minute glucose ≥ 200 mg/dL b. HbA1c ≥ 5.7 c. Index60 ≥ 1.4 d. Diabetes Prevention Trial-Type 1 Risk Score (DPTRS) ≥ 7.4
5. Females of childbearing potential must agree to use abstinence or an effective birth control through the treatment period.(
6. Males able to father children, must agree to use abstinence or an effective birth control during the treatment period.
7. Subjects who are Epstein-Barr virus (EBV) seronegative at screening must be EBV Polymerase chain reaction (PCR) negative within 30 days of randomization and may not have had signs or symptoms of an EBV compatible illness lasting longer than 7 days within 30 days of randomization
8. Be at least 4 weeks from last live immunization
9. Be willing to forgo live vaccines through and 3 months after study drug treatment period
10. Be up to date on all recommended vaccinations based on age of subject and willing to receive killed influenza vaccine when available for current or upcoming season.
11. If prior treatment with active study agent from previous clinical trial, approval of medical monitor and investigator that such prior treatment does not impact risk for current study.
12. Subjects who have met all above criteria must have the qualifying oral glucose tolerance test (OGTT) within 7 weeks (52 days) of randomization and baseline visit.

Exclusion Criteria:

Potential participants must not meet any of the following exclusion criteria:

* 1. Be immunodeficient or have clinically significant chronic lymphopenia: (Leukopenia (< 3,000 leukocytes /μL), neutropenia (<1,500 neutrophils/μL), lymphopenia (<800 lymphocytes/μL), or thrombocytopenia (<100,000 platelets/μL).

  2. Have active signs or symptoms of acute infection at the time of randomization including Sars-Cov2.

  3. Have evidence of prior or current tuberculosis infection as assessed interferon gamma release assay (QuantiFERON).

  4. Be currently pregnant or lactating, or anticipate getting pregnant within the study period

  5. Require chronic use of other immunosuppressive agents including use of inhaled, intranasal, or systemic steroids

  6. Have evidence of current or past HIV, Hepatitis B, histoplasmosis, coccidioidomycosis, or current Hepatitis C infection.

  7. Have any complicating medical issues or abnormal clinical laboratory results that may interfere with study conduct, or cause increased risk to include pre-existing pulmonary, GI, renal, cardio-vascular disease, neurological disease (i.e. demyelinating disease), psychiatric disease or blood count abnormalities. Note pre-existing treated celiac or thyroid disease are not exclusionary diagnoses.

  8. Have a history of malignancies other than of skin

  9. Evidence of liver dysfunction with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 2 times the upper limits of normal

  10. Evidence of renal dysfunction with creatinine greater than 1.5 times the upper limit of normal for age and sex.

  11. Known history of congestive heart failure or left ventricular dysfunction.

  12. Vaccination with a live virus within the last 4 weeks

  13. Current or ongoing use of non-insulin pharmaceuticals that affect glycemic control within 30 days of screening (see section 4.5 for list of exclusionary pharmaceuticals).

  14. Active participation in another intervention study in the previous 30 days

  15. Known allergy to Anti-TNFα or latex.

  16. Any condition that in the investigator's opinion may adversely affect study participation or may compromise the study results

  17. Previously diagnosed with T1D according to American Diabetes Association (ADA) criteria

Ages: 3 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the elapsed time from random treatment assignment to the development of diabetes (T1D) or time of last contact among those randomized | 6 years
  The primary outcome is the elapsed time from random treatment assignment to the development of diabetes (T1D) or time of last contact among those randomized

CONTACTS AND LOCATIONS:
Overall Officials: Carla Greenbaum, MD, Study Chair — Type 1 Diabetes TrialNet

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available at the National Institute of Diabetes Digestive and Kidney Diseases (NIDDK) Central Repository
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- See also: TrialNet Public Website — http://www.trialnet.org/